CLINICAL TRIAL: NCT05190302
Title: Determination of the Sensitivity, Specificity and Receiver Operating Characteristic of Nerve Stimulation Receptor as a Decision-making Tool During Ultrasound Guided Peripheral Nerve Block - a Feasibility Study (StimUtile - Phase I)
Brief Title: Determination of the Sensitivity, Specificity & Receiver Operating Characteristic of Nerve Stimulation Receptor as a Decision-making Tool During US Guided PNB
Status: Terminated | Type: Observational
Why Stopped: During the course of the year, we were able to answer our faisability question.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 21.294
Record Dates: First submitted 2021-12-21; First posted 2022-01-13 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Nerve Block
Keywords: Neurostimulation; Neuropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phase I - Patients undergoing regional anesthesia with a block allowing a neurostimulation.: The investigators propose to conduct a single-blind, prospective observational study on all eligible patients undergoing regional anesthesia with a peripheral nerve block allowing a neurostimulation.

SUMMARY:
Although the superiority of ultrasound guidance over neurostimulation (NS) has been demonstrated, it has its limits, namely when used for a deeper block (device limits) or if used by a less experienced operator (ability to recognize structures, to correctly position the needle). In addition, its use has failed to consistently prevent intra-neural injection.

The question of the usefulness of NS in addition to ultrasound is therefore still relevant. A great geographical disparity exists in the habits of nerve localization. The reluctance to use NS stems mainly from doubts about its effectiveness. The threshold used to consider that the needle is sufficiently close to the nerve and the one used to exclude an intraneural injection have been disputed in several studies. Another weakness of studies concerning NS since the advent of ultrasound guidance is the impossibility of generalizing the results. All clinical studies were performed in an academic setting, and a large majority of them specify that the blocks were performed by - or supervised by - regional anesthesia experts.

The only study that attempted to determine the sensitivity of NS used ultrasound as a gold standard. The choice of the ultrasound position as the gold standard is debatable, since it is dependent of the operator. The clinical success of nerve blocks would be a better standard.

No study to date has made it possible to calculate the specificity and sensitivity of NS in addition to ultrasound guidance, and therefore, to obtain the positive and negative predictive values of the technique. Obtaining these values could allow each clinical setting or individual to determine the contribution of NS to their rate of success, as a modest increase in the success rate or a minimal decrease in the risk of neuropathy would be clinically significant.

The hypothesis is that the sensitivity and specificity of NS justifies its use in combination with ultrasound guidance in most settings, but that the gain in efficiency varies depending on the context (for example depending on the local success rate).

To determine the required sample size to test this hypothesis and plan for a definitive study on the question, the investigators need to know what is the local failure rate (incidence of studied event) and what could be the possible rate of patient enrollment.

This preliminary, feasibility study will aim to confirm that the local failure rate is compatible with the 5% rate observed in the literature.

DETAILED DESCRIPTION:
This study is a single-blind, prospective observational study including patients 18 years and older, undergoing regional anesthesia with a peripheral nerve block allowing a neurostimulation.

This study is a phase I of a three-phases program to determine the feasibility of a larger study and to refine the sample size calculation for the phase II, currently estimated at 2,140 patients. The phase II would aim to determine whether neurostimulation improves the success rate for ultrasound-guided nerve block. If the first two phases are successful, a phase III, multicentric, will be considered to determine the usefulness of neurostimulation in addition to guidance ultrasound for the prevention of nerve complications from peripheral regional anesthesia.

The primary objective of Phase I is to determine the local failure rate of ultrasound-guided nerve block techniques, in order to refine the sample size calculation.Since patients from phase I will be included in the analysis for phase II, the study protocol and collected data will be the same as for the subsequent phases.

The secondary objectives of Phase I are to:

* Determine if a recruitment rate of three patients per day is possible
* Evaluate the staff time required for each patient recruited
* Determine if the data can be obtained completely and reliably.

The blocks included in this study are:

* Brachial plexus block by interscalene approach
* Brachial plexus block by supraclavicular approach
* Brachial plexus block by infraclavicular approach
* Specific brachial branch plexus blocks in mid-humeral, elbow or proximal part of the forearm
* Femoral nerve block by inguinal approach
* Obturator nerve block
* Sciatic nerve block by infra-gluteal approach
* Sciatic nerve block by popliteal approach

The type of block will be left to the discretion of the anesthesiologist, but must imperatively be done under real-time ultrasound guidance. Co-analgesia (Acetaminophen, Celecoxib, etc.) and sedation may be administered depending on the decisions of the treating anesthesiologist. The positioning will be left to the choice of the operator.

After the desinfection of the skin, the ultrasound will be used during the block to guide and to obtain an image of the needle point near the target (root/cord/nerve)

When the anesthesiologist is satisfied of the position, the assistant will start the neurostimulation with an intensity of 1.0 mA (Pajunk MultiStim Sensor, Germany). The intensity will be decreased to determine the value where all distal muscular response disappears. This intensity will be noted. However, the anesthesiologist will not be aware of the motor response (threshold) unless the value is below 0.3 mA. In this case, the anesthesiologist will be free to decide whether the needle should be repositionned.

Should the anesthesiologist decide to reposition the needle, the neurostimulation process will be repeated.

The anesthesiologist may then inject a small volume of dextrose 5% solution with a pressure limiting device (Nerve guard, Pajunk) to confirm adequate distribution of the solution and adequate pressure.

If unsatisfied, the anesthesiologist can again reposition the needle and repeat the neurostimulation process.Injection of dextrose prior to stimulation will be noted by the investigation team because that may change the neurostimulation profile of the targeted nerve.

Prior to the final injection of the local anesthetic, a intra-neural test dose of 3 mL will be injected to try to identify an "early block" which could underline an intra-neural positionning of the needle. In absence of immediate effect, the injection can be done according to the usual approach of the treating team.

Once in the OR, the usual maneuvers will be done to determine the efficacy of the block.

The success of the block will be documented at 30 minutes after the bloc (T1), just before the beginning of the intervention (T2) as well as at the end of the anesthesia (T3).

A phone call will be done 24 hours post-op if a unique injection was given or 24 hours after the end of the perfusion, if given in continuous infusion via catheter, to collect any complications related to the peripheral block.

Data analysis

A sample size of 200 patients was determined for phase I of this study in order to meet the primary objective.

Descriptive statistics on data relating to the research process will help determine the feasibility of the study and the resources involved.

A simple incidence calculation with confidence intervals will determine the block failure rate of the peripheral ultrasound-guided nerve block.

The average recruitment rate per day will be calculated, with confidence intervals.

The staff time required for each patient with confidence intervals will be calculated.

The clinical data will be analyzed in an exploratory manner. The data will be analyzed according to the effectiveness of the block (complete / incomplete) in relation to the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

A preliminary ROC curve will be determined by modifying the minimum threshold value and noting the effect on the neurostimulation sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years and older, undergoing regional anesthesia with a peripheral nerve block allowing a neurostimulation.

Exclusion Criteria:

* Contraindications to a peripheral nerve block
* Risk of severe intoxication to local anesthesia
* Peripheral nerve block in an area not allowing neurostimulation due to absence of motor fibers (for example, adductor canal block)
* Patient refusal
* Patient unable to communicate with the health or research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years and older, undergoing regional anesthesia with a peripheral nerve block allowing a neurostimulation.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound-guided peripheral nerve block failure rate | At the end of the Phase I study, with an estimated duration of 4 months
  A block will be considered a success if the patient has complete motor and sensory block, no pain or discomfort in the target area requiring the addition of any analgesic agent during surgery. A conversion to unplanned general anesthesia would constitute a failure of the block.

SECONDARY OUTCOMES:
Recruitment rate | At the end of the Phase I study, with an estimated duration of 4 months
  The number of patients recruited each day.
Recruitment time | At the end of the Phase I study, with an estimated duration of 4 months
  Time required to recruit each patient.
Completeness of the data collected | At the end of the Phase I study, with an estimated duration of 4 months
  Percentage of patients with complete case reports forms.
Reliability of the data collected | At the end of the Phase I study, with an estimated duration of 4 months
  Average percentage of data collected/patient.
Incidence of breach in protocol | At the end of the Phase I study, with an estimated duration of 4 months
  The rate of protocol deviations occurring in the study population over the time of the study.
Losses to follow-up | At the end of the Phase I study, with an estimated duration of 4 months
  Number of patients who are not contacted or who withdraw from the study before the 24h follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Garneau, MD, FRCPC, Principal Investigator — Centre Hospitalier de l'Université de Montreal - CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No